CLINICAL TRIAL: NCT04456062
Title: Using Caring Contacts to Reduce Psychiatric Morbidity Following Hospitalization During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ayal Schaffer, Staff Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1804
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Psychiatric Hospitalization
Keywords: Caring Contacts; Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caring Contacts Group (Experimental)
  Interventions: Other: Caring Contacts
- Standard Treatment Group (No Intervention)

INTERVENTIONS:
Other: Caring Contacts — Caring Contacts are brief email communications sent to the patient post-discharge. They convey messages of hope, support, promote a sense of belonging, and provide information on resources for care. They are not written uniquely for each patient but are purposefully crafted to intervene on those specific vulnerabilities that form the core of many patients' experiences with intense emotional distress and suicidal thoughts.
  Arms: Caring Contacts Group

SUMMARY:
Subjects will be recently discharged patients from Sunnybrook Inpatient Psychiatry Unit. Subjects will be randomized in a 1:1 ratio to either the Caring Contact intervention or usual care. 75 subjects will be enrolled in each arm. In additional to usual discharge-related care, subjects in the caring contact group will receive brief emails that convey a message of hope and provide resources. These emails will be sent on days 4, 21, and 56 post-discharge. The specific content of these emails will be pre-determined varying slightly by time point. In contrast, the control group will only receive usual discharge-related care, including discharge planning and also a sheet of resources normally provided to patients. A widely used and validated measure will be employed to assess depression and anxiety symptoms. The 25-item self-report Hopkins Symptom Checklist will be emailed to all subjects at baseline, day 4, 21, and 56 post-discharge, along with the Caring Contact communication. It is hypothesized that there will be a significantly greater reduction in mental health symptoms among patients receiving Caring Contacts compared to those who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Inpatient status in Sunnybrook Inpatient Psychiatry Unit at time of recruitment
* Have an email or mailing address
* Ability to read and understand English
* The ability to understand and comply with the requirements of the study and capable of providing informed consent

Exclusion Criteria:

* A primary Major Neurocognitive Disorder diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Baseline, day 4, day 21, day 56 post-discharge
  The HSCL-25 is a widely-used and validated self-report questionnaire using a Likert scale to measure symptoms of anxiety and depression. Change scores in anxiety and depression will be used to assess effectiveness of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Schaffer, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Rosalie Steinberg, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Holman S, Steinberg R, Sinyor M, Lane H, Starritt K, Kennedy SH, Niederkrotenthaler T, Zaretsky A, Castel S, Schaffer A. Caring Contacts to Reduce Psychiatric Morbidity Following Hospitalization During the COVID-19 Pandemic: A Pilot Randomized Controlled Trial. Can J Psychiatry. 2023 Mar;68(3):152-162. doi: 10.1177/07067437221121111. Epub 2022 Aug 22. PMID 35996823